CLINICAL TRIAL: NCT04126395
Title: An Explorative Retrospective Video-analysis of the Motor Development of Children With Developmental Coordination Disorder Before the Age of Two
Brief Title: An Explorative RVA of the Motor Development of Children With DCD <2y
Acronym: RVA_DCD
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-05716
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Developmental Coordination Disorder; Autism Spectrum Disorder
Keywords: motor development; baby; infant; motor milestones; crawling; independent walking
MeSH Terms: conditions — Motor Skills Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: This groups consists of children now aged 6-12y:
  * Without a medical diagnosis possibly influencing motor development
  * Without motor problems (M-ABC-2 and DCD-Q)
  * Without social reponsiveness problems (SRS-2)
  Interventions: Diagnostic Test: Movement Assessment Battery for Children 2(M-ABC-2); Diagnostic Test: Developmental Coordination Disorder - Questionnaire (DCD-Q); Diagnostic Test: Social Responsiveness Scale 2 (SRS-2); Other: Retrospective Video Analysis
- Developmental Coordination Disorder: This groups consists of children now aged 6-12y:
  * With a multidisciplinary diagnosis of DCD
  * With motor problems (M-ABC-2 and DCD-Q)
  Interventions: Diagnostic Test: Movement Assessment Battery for Children 2(M-ABC-2); Diagnostic Test: Developmental Coordination Disorder - Questionnaire (DCD-Q); Diagnostic Test: Social Responsiveness Scale 2 (SRS-2); Other: Retrospective Video Analysis
- Developmental Coordination Disorder + Autism Spectrum Disorder: This groups consists of children now aged 6-12y:
  * With a multidisciplinary diagnosis of DCD
  * With motor problems (M-ABC-2 and DCD-Q)
  * With social responsiveness problems (SRS-2)
  Interventions: Diagnostic Test: Movement Assessment Battery for Children 2(M-ABC-2); Diagnostic Test: Developmental Coordination Disorder - Questionnaire (DCD-Q); Diagnostic Test: Social Responsiveness Scale 2 (SRS-2); Other: Retrospective Video Analysis

INTERVENTIONS:
Diagnostic Test: Movement Assessment Battery for Children 2(M-ABC-2) — The M-ABC-2 is a motor performance test for children aged 3 trough 16 years of age. We will use Dutch-Flemish norms.
Diagnostic Test: Developmental Coordination Disorder - Questionnaire (DCD-Q) — The DCD-Q is a brief parent questionnaire designed to screen for the presence of DCD in children aged 5 trough 15 years of age. We will use Dutch norms.
Diagnostic Test: Social Responsiveness Scale 2 (SRS-2) — The SRS-2 is a parent questionnaire designed to identify social impairments associated with ASD in children 4 trough 18 years of age. We will used Dutch norms.
Other: Retrospective Video Analysis — Retrospective video analysis will be used to explore motor development in children with DCD, DCD+ASD and controls.

SUMMARY:
This study compares motor development in three groups of infants (controls, DCD, DCD+ASD) before the age of 2 years using retrospective video analysis of infants in home video contexts.

ELIGIBILITY:
CONTROLS:

Inclusion Criteria:

* Availability of video material of the child before the age of 2.
* No indication of DCD (as measured by M-ABC-2 Pc>16 and DCD-Q)
* No indication of ASD (as measured by SRS-2 T-score ≤60 )

Exclusion Criteria:

* Medical diagnosis possibly influencing motor development (DCD, ASD, ADHD, CP, ect)
* Severe ilnesses in the early Developmental period (0-2y) which may have influenced the development (f.e. CVA, cancer, severe traumas,...)
* Prolonged admission to the hospital (≥ 3 weeks) in the early Developmental period (0-2y)

DCD GROUP:

Inclusion criteria:

* Availability of video material of the child before the age of 2.
* Formal diagnosis of DCD provided by multidisciplinary team in Flanders
* Indication of DCD (as measured by M-ABC-2 Pc≤16 and DCD-Q)

Exclusion Criteria:

* Other medical diagnosis possibly influencing motor development (ASD, ADHD, CP, ect)
* Severe ilnesses in the early Developmental period (0-2y) which may have influenced the development (f.e. CVA, cancer, severe traumas,...)
* Prolonged admission to the hospital (≥ 3 weeks) in the early Developmental period (0-2y)

DCD+ASD GROUP:

Inclusion criteria:

* Availability of video material of the child before the age of 2.
* Formal diagnosis of DCD and ASD provided by multidisciplinary team in Flanders
* Indication of DCD (as measured by M-ABC-2 Pc≤16 and DCD-Q)
* Indication of ASD (as measured by SRS-2 T-score >60 )

Exclusion Criteria:

* Other medical diagnosis possibly influencing motor development (ADHD, CP, ect.)
* Severe ilnesses in the early Developmental period (0-2y) which may have influenced the development (f.e. CVA, cancer, severe traumas,...)
* Prolonged admission to the hospital (≥ 3 weeks) in the early Developmental period (0-2y)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Observable Movement Quality Scale | 0-2years
  The OMQ is a standardized 15-item observational scale to asses the movement quality. A maximum of two 5-minute compilations are assembled per child per age-category (6-12 months, 12-18 monhts, 18-24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Van Waelvelde, Dr., Principal Investigator — University Ghent
Locations (2):
- Ghent University, Ghent, Belgium
- UBC, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No